CLINICAL TRIAL: NCT05982860
Title: Evaluation of the Effects of the MIND Diet on Oxidative Stress, Inflammation and Neurodegenerative Risk Biomarkers in American Football Players
Brief Title: The Effects of the MIND Diet on Oxidative Stress, Inflammation and Neurodegenerative Risk Biomarkers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bartu Eren Güneşliol (Other)
Collaborators: Gazi University (Other)
Responsible Party: Sponsor-Investigator, Bartu Eren Güneşliol, Research Assistant, Duzce University
Organization: Duzce University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: BARTU 01
Record Dates: First submitted 2023-08-01; First posted 2023-08-09 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Neurodegeneration; Inflammation; Oxidative Stress; Diet, Healthy; Diet Habit; Nutrition, Healthy
Keywords: MIND diet; sports nutrition; Dietary habits; Neurodegeneration; Inflammation; Oxidative stress
MeSH Terms: conditions — Nerve Degeneration; Inflammation; Feeding Behavior

STUDY DESIGN:
Intervention Model Description: This study was planned as a randomized controlled trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (n:18) (No Intervention): Players in this group will not be given any nutritional advice/intervention. They will maintain their usual eating habits.
- MIND diet (n:18) (Experimental): Players in this group will be asked to include the food groups in the MIND diet in their diet in accordance with their consumption frequency. As a result of the interviews with the coaches and experienced athletes, it was learned that the majority of the athletes did not consume the foods such as wine, berries, and fish included in the MIND diet template. Therefore, these foods, which are the main components of the MIND diet, will be provided by the researcher/project in accordance with the recommended frequencies. However, since wine consumption is not frequently preferred in our country due to religious and socio-cultural reasons, ''hardaliye'', a fermented grape juice (100 mL/day), which is easy to consume and has similar nutritional values to wine (resveratrol and ORAC), will be provided. Berries will be supplied in 2 portions/week, and fish (tons) in 1 portion/week.
  Interventions: Behavioral: MIND diet

INTERVENTIONS:
Behavioral: MIND diet — Mediterranean-DASH Intervention for Neurodegenerative Delay (MIND) diet has been established by Morris et al. (2015) to improve brain health, and reduce the risk or slow progression of neurodegenerative diseases. In this diet model, which is similar to the Mediterranean diet, the diet score changes according to the frequency of consumption of some foods. The more consumption of foods such as green leafy vegetables, other vegetables, berries, nuts, whole grains, fish (not fried), beans, poultry (not fried), and the limited consumption of butter/margarine, cheese, red meat and products, fast fried foods, and pastries & sweets ensure more score. Also, regular consumption of wine (1 glass/d) and using olive oil as primary oil in meals increases the score. Berries, fish, and hardaliye (instead of wine) will be supplied to players as well as recommendations for consumption frequencies of food components in MIND diet to increase total score.
  Arms: MIND diet (n:18)

SUMMARY:
American football is a high-contact sport, also known as a collision sport. American football players are exposed to various magnitudes and frequencies of head impacts throughout the season. Accordingly, during the American football season, there is an increase in biomarkers that may be associated with brain damage and the risk of developing neurodegenerative diseases later in life. In addition, oxidative stress and inflammation can also increase in athletes during the American football season. This study was planned with the thought that the MIND diet, which is beneficial for brain health with its antioxidant and anti-inflammatory effects, may have positive effects on oxidative stress, inflammation and neurodegenerative risk biomarkers in American football players.

The goal of this clinical trial is to examine the effects of the MIND diet on oxidative stress, inflammation and neurodegenerative risk biomarkers in American football players. The main question it aims to answer are:

• [Question] Does the MIND diet lowers or reduce the levels of oxidative stress, inflammation and neurodegenerative risk biomarkers in American football players?

Participants will be randomized into 2 groups MIND diet and control group. The current diet of the players in the control group will not be interfered with during the competition period, but the current nutrition of the players in the MIND diet group will be adapted to the MIND diet according to the food groups in the MIND diet components and their consumption frequencies.

The players in the MIND diet group will be asked to include the food groups in the MIND diet in their diet in accordance with their consumption frequency.

Researchers will compare the MIND diet and control groups to see if the MIND diet improves oxidative stress, inflammation and neurodegenerative risk biomarkers.

DETAILED DESCRIPTION:
American football is one of the contact sports with the highest risk in terms of exposure to repeated head impacts and the formation of neurodegenerative diseases that negatively affect the quality of life in the later stage of life. According to studies conducted in recent years, these athletes have a high risk of developing neurodegenerative diseases such as Alzheimer's, amyotrophic lateral sclerosis (ALS) and chronic traumatic encephalopathy (CTE) later in life. It has been reported that there are increases in the levels of oxidative stress, inflammation and neurodegenerative risk biomarkers and that some other biomarkers (such as BDNF, zonulin, telomere length, etc.) that may be associated with these may be adversely affected in American football players. It is necessary to develop new approaches to determine the preventive factors against the risk of neurodegenerative diseases that may occur in the later years of life due to contact sports such as American football. The Mediterranean-DASH Intervention for Neurodegenerative Delay (MIND) diet has antioxidant (vitamins, flavonoids, phytosterols, minerals, terpenes and phenols) and anti-inflammatory (oleic acid, polyphenols and unsaturated fatty acids) properties that are thought to be effective in improving oxidative stress, inflammation and neurodegenerative risk biomarkers. The MIND diet can also reduce intestinal permeability with its abundant fiber content (prebiotic effect). It has been reported that the supplementation of some nutrients (docosahexaenoic acid, eicosapentaenoic acid, etc.) that have an important place in the composition of the MIND diet in this group of athletes has a positive effect on some of these biomarkers. However, the studies in the literature are limited, and there is no study involving the MIND diet in American football players. This study was planned considering that the MIND diet may have positive effects on oxidative stress, inflammation, and neurodegenerative risk biomarkers in American football players, who are exposed to repetitive head impacts as a nature of this contact sport.

American football players playing in the pro league will be included in this study. The sample size was calculated using the G*Power V. 3.1.9.6 program. This study will include two groups and two measurements. Accordingly, a total of 30 athletes, 15 in each group, with 95% confidence (1-α), 95% test power (1-β) and f=0.6 effect size; with 80% confidence (1-α), 80% test power (1-β) and f=0.6 effect size, a total of 20 athletes, 10 in each group, should be included.

At the beginning of the research, a face-to-face questionnaire will be used to question the athletes' American football history and player positions, socio-demographics, general health and nutritional habits. Before the start of the study, a 7-day food consumption record will be taken from the athletes. MIND scores will be questioned before the study and every week till the end of the study according to the frequency of food consumption in the MIND composition scale. It will be used to assess participants' adherence to the MIND diet. Accordingly, the MIND diet components include ten food groups (green leafy vegetables, other vegetables, nuts, berries, bean types, whole grains, seafood, poultry, olive oil, and wine) that are healthy for the brain. There are also five food groups (red meat, butter and margarine, cheese, pastries and sweets and fried / fast food / fast food) that are considered unhealthy. Frequencies of food consumption (daily, weekly, monthly) are questioned according to whether these 10 food groups specified in the template are preferred based on portion and meal or as primary, and as a result, scoring is made as 0, 0.5 and 1 points for each food group. The highest score is 15 points. Because the MIND diet template does not have specific scores for diet adherence, below the median score (7.5) will be considered low adherence. According to the MIND diet composition scale, those with a MIND diet score of <7.5 points will be included in the study, while those with a score of ≥7.5 will be excluded from the study. At the beginning of the study, body composition measurements (anthropometric measurements and bioelectrical impedance analysis) will be taken from the athletes along with the Pittsburgh sleep quality index scale scores, diet inflammatory index, and the World Health Organization quality of life scale-short form. Oxidative stress, inflammation, neurodegenerative risk and other associated biomarkers will be analyzed in blood samples.

Athletes will be randomized into two groups; MIND diet and control group. The players in the control group will sustain their habitual nutrition, while the current nutrition of the players in the MIND diet group will be adapted to the MIND diet according to the food groups in the MIND diet components and their consumption frequencies. In this context, the players will be informed about the general characteristics of the MIND diet and its importance in terms of their health. To help the participants in this regard, information will be given about the changes in the size and amount of foods and their portions in general with the "Meal and Food Photo Catalogue". As a result of the interviews with the coaches and experienced players, it was learned that the majority of the players did not consume/can't access the foods such as wine, berries, and fish included in the MIND diet template. Therefore, these foods, which are the main components of the MIND diet, will be provided by the researcher/project by the recommended frequencies. However, since wine consumption is not frequently preferred in our country due to religious and socio-cultural reasons, ''hardaliye'' (100 mL/day), which is easy to consume and has similar nutritional values to wine (resveratrol and ORAC), will be provided. Red forest fruits will be supplied in 2 portions/week, and fish (tons) in 1 portion/week. Before the study, participants assigned to the MIND diet group were provided with brochures, information, presentations, etc. so that they could adapt to the MIND diet. Participants in this group will be supported during the study period to increase their adherence to the MIND diet with information and suggestions via phone, mail, WhatsApp groups, etc. Those in the MIND diet group with an overall mean MIND score of <7.5 at mid- or end-of-study will be excluded from the study. Athletes in the control group with an overall mean MIND score of ≥7.5 at the mid- or end-of-study will be excluded from the study. Since all teams will participate in the same number of competitions and the group matches will last approximately nine weeks, the follow-up time has been determined as nine weeks. At the end of the nine-week follow-up, all parameters evaluated at the beginning of the study will be taken again, and the last values will be compared with the previous values.

ELIGIBILITY:
Inclusion Criteria:

* Having played American football for at least 2 years
* ≥18 years old
* Having had a MIND diet score of < 7.5 points
* Not having any family or cohabitants following the MIND diet
* Providing written informed consent

Exclusion Criteria:

* <18 years old
* Having had a MIND diet score of ≥7.5 points
* History of concussion diagnosed in the last 6 months
* use of anti-inflammatory or antioxidant drugs (>20 days)
* food allergy
* A state of injury that is unable to carry out the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Since only men play American football, our study is based on male gender.
Enrollment: 24 (Actual)
Dates: Start 2023-06-23 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2025-06-05 (Actual)

PRIMARY OUTCOMES:
Tau protein | Before and after the 9-week research.
  A biomarker associated with disruption of the blood-brain barrier, neuroinflammation and brain damage caused by repetitive head impact or concussion occurring during American football games and considered an indicator of neurodegenerative risk.
NfL (Neurofilament light polypeptide) | Before and after the 9-week research.
  A biomarker associated with disruption of the blood-brain barrier, neuroinflammation and brain damage caused by repetitive head impact or concussion occurring during American football games and considered an indicator of neurodegenerative risk.
S100B protein | Before and after the 9-week research.
  A biomarker associated with disruption of the blood-brain barrier, neuroinflammation and brain damage caused by repetitive head impact or concussion occurring during American football games and considered an indicator of neurodegenerative risk.
BDNF (Brain Derived Neurotrophic Factor) | Before and after the 9-week research.
  A biomarker associated with an important role in reducing neurodegenerative risk and in cellular events occurring in restorative processes against damage that may lead to oxidative stress and neuroinflammation in contact sports such as American football.
Telomere | Before and after the 9-week research.
  Due to increased oxidative stress and inflammation, the erosion of telomeres, a biomarker of aging, may occur more rapidly. Damaged mitochondria in American football players can trigger an increase in oxidative stress and inflammation levels, which are the most important triggers of the mechanisms of neurodegenerative disorders, and lead to cell death. Telomere shortening is associated with premature cellular senescence and cell death and is thought to be a biomarker for neurodegenerative damage at the cellular level.
Zonulin | Before and after the 9-week research.
  Low serum zonulin levels appear to be a biomarker for increased intestinal permeability and disruption of gastrointestinal barrier integrity. Increased intestinal permeability and disruption of intestinal barrier integrity may also increase already existing neuroinflammation by increasing inflammation.
NOX2 (NADPH oxidase) | Before and after the 9-week research.
  A biomarker of oxidative stress. American football training and competition periods can cause excessive free radical production and cause oxidative stress.
8-OHdG (8- hydroxy-2-deoxyguanosine) | Before and after the 9-week research.
  A biomarker of oxidative stress. American football training and competition periods can cause excessive free radical production and cause oxidative stress.
F2-isoprostanes (F2-isoPs) | Before and after the 9-week research.
  A biomarker of oxidative stress. American football training and competition periods can cause excessive free radical production and cause oxidative stress.
hs-CRP (High-sensitivity C-reactive protein) | Before and after the 9-week research.
  A biomarker of inflammation. The concentrations of inflammatory biomarkers can increase during American football training and competition periods.
IL-6 (Interleukin 6) | Before and after the 9-week research.
  A biomarker of inflammation. The concentrations of inflammatory biomarkers can increase during American football training and competition periods.
TNF-α (Tumor necrosis factor alpha) | Before and after the 9-week research.
  A biomarker of inflammation. The concentrations of inflammatory biomarkers can increase during American football training and competition periods.

SECONDARY OUTCOMES:
Sleep quality score | Before and after the 9-week research.
  The Pittsburgh Sleep Quality Index (PSQI) will be used to assess sleep quality.
Quality of life score | Before and after the 9-week research.
  The quality of life will be assessed via the questionnaire of The World Health Organization quality of life (WHOQOL).
Dietary inflammatory index (DII) score | Before and after the 9-week research.
  Dietary inflammatory index will be calculated based on formula originally developed by Shivappa et al. (2014).

CONTACTS AND LOCATIONS:
Overall Officials: Bartu Gunesliol, Master, Principal Investigator — Duzce University; Nilufer Tek, PhD, Principal Investigator — Gazi University; Asiye Dikmen, PhD, Principal Investigator — Gazi University
Locations (1):
- Duzce University, Düzce, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
It is considered that the scientific outputs of the study could be shared upon request without personal data. Any participants' private data will never be shared. Personal private data protection law will be complied with.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: It is expected that access to the scientific outputs of this research will be provided from 2025 and will be open until 2028.
Access Criteria: It is planned to be accessible only to international academic staff and researchers.